CLINICAL TRIAL: NCT04065841
Title: A Randomized, Double-blind, Parallel-group, Multicenter Study to Assess Efficacy, Safety, and Tolerability of Oral Tropifexor (LJN452) & Licogliflozin (LIK066) Combination Therapy and Each Monotherapy, Compared With Placebo for Treatment of Adult Patients With Nonalcoholic Steatohepatitis (NASH) and Liver Fibrosis.(ELIVATE)
Brief Title: Efficacy, Safety and Tolerability of the Combination of Tropifexor & Licogliflozin and Each Monotherapy, Compared With Placebo in Adult Patients With NASH and Liver Fibrosis.
Acronym: ELIVATE
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The sponsor made a business decision to stop development of the trial drugs. The decision to stop the trial early was not because of any safety concerns.
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLJN452D12201C; 2019-002324-32 (EudraCT Number)
Record Dates: First submitted 2019-08-19; First posted 2019-08-22 (Actual); Results first posted 2023-12-26 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Non Alcoholic Steatohepatitis (NASH)
Keywords: NASH; Non alcoholic steatohepatitis; Tropifexor; LJN452; Licogliflozin; LIK066; Placebo
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — tropifexor; licogliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Arm A: combination therapy (Experimental): Combination therapy arm: tropifexor 140 mcg capsule + licogliflozin 30 mg tablet, once daily orally
  Interventions: Drug: Tropifexor; Drug: Licogliflozin
- Arm B: tropifexor monotherapy (Experimental): Tropifexor monotherapy arm: tropifexor 140 mcg capsule (+ placebo matching licogliflozin tablet), once daily orally
  Interventions: Drug: Tropifexor
- Arm C: licogliflozin monotherapy (Experimental): Licogliflozin monotherapy arm: licogliflozin 30 mg tablet (+ placebo matching tropifexor capsule), once daily orally
  Interventions: Drug: Licogliflozin
- Arm D: Placebo (Placebo Comparator): Placebo arm: placebo matching tropifexor capsule + placebo matching licogliflozin tablet, once daily
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Tropifexor — 100mcg+30mcg+10mcg capsules of tropifexor taken orally every day until the 140 mcg capsule of tropifexor taken orally every day is produced, then patients will switch to the single 140mcg capsule taken orally every day
  Other Names: LJN452
  Arms: Arm A: combination therapy; Arm B: tropifexor monotherapy
Drug: Licogliflozin — 30mg tablet of licoglifozin taken orally every day
  Other Names: LIK066
  Arms: Arm A: combination therapy; Arm C: licogliflozin monotherapy
Other: Placebo — licogliflozin placebo + tropifexor placebo
  Arms: Arm D: Placebo

SUMMARY:
Randomized, double-blind, parallel-group, multicenter study to assess efficacy, safety, and tolerability of oral tropifexor & licogliflozin combination therapy and each monotherapy, compared with placebo for treatment of adult patients with nonalcoholic steatohepatitis (NASH) and liver fibrosis.

DETAILED DESCRIPTION:
The study consisted of 1) a screening period, 2) a treatment period starting from randomization on Day 0 and running to Week 48, and 3) a follow-up period of 4 weeks after the last dose of study treatment. The study duration from first dose of study medication was 52 weeks.

ELIGIBILITY:
Inclusion Criteria:

Presence of NASH with fibrosis confirmed by central reader's evaluation of liver biopsy obtained no more than 6 months before randomization as demonstrated by the following:

1. NASH using NAFLD Activity Score (NAS) ≥ 4 with at least 1 point each in inflammation and ballooning and
2. Fibrosis stage 2 or 3 using NASH CRN fibrosis criteria

Exclusion Criteria:

* Type 1 diabetes mellitus
* Uncontrolled type 2 diabetes defined as glycated hemoglobin (HbA1c) ≥ 9.0% at screening
* HbA1c < 6.5% at screening in Type 2 diabetics currently treated with insulin or sulfonylureas
* Clinical evidence of liver impairment as defined by the presence of any of the following abnormalities:

  * Platelet count < LLN (see Central laboratory manual).
  * Serum albumin < LLN (see Central laboratory manual).
  * International Normalized Ratio (INR) > ULN (see Central laboratory manual).
  * ALT or AST > 5× ULN (confirmed by 2 values during screening).
  * Total bilirubin > ULN (see Central laboratory manual) (confirmed by 2 values during screening), including Gilbert's syndrome.
  * Alkaline phosphatase > 300 IU/L (confirmed by 2 values during screening).
  * History of esophageal varices, ascites or hepatic encephalopathy
  * Splenomegaly
  * MELD score >12

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 234 (Actual)
Dates: Start 2019-12-30 (Actual); Primary Completion 2022-10-27 (Actual); Study Completion 2022-10-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (75):
- United States (28):
  - Gut PC Digestive Health Specialist, Dothan, Alabama
  - Southern California Research Center, Coronado, California
  - Velocity Clinical Trials, Los Angeles, California
  - California Liver Research Institute, Pasadena, California
  - Medical Associates Research Group, San Diego, California
  - San fernando Valley Health Institute, Van Nuys, California
  - Island View Gastroenterology Associates, Ventura, California
  - Integrity Clinical Rsh LLC, Doral, Florida
  - Galenus Group, Lehigh Acres, Florida
  - Genoma Research Group Inc, Miami, Florida
  - Digestive Res Alliance of Michiana, South Bend, Indiana
  - Southern Therapy and Adv Res LLC, Jackson, Mississippi
  - Clinical Research Professionals Inc, Chesterfield, Missouri
  - Southwest Gastroenterology Associates, Albuquerque, New Mexico
  - Northwell Health, Manhasset, New York
  - Clinical Trials Of America LLC, Lenoir, North Carolina
  - Diabetes And Endocrinology Conslt, Morehead City, North Carolina
  - Options Health Research, Tulsa, Oklahoma
  - Prisma Health, Greenville, South Carolina
  - Digestive Disease Research, Greenwood, South Carolina
  - Palmetto Clinical Research, Summerville, South Carolina
  - Summit Medical Care, Hermitage, Tennessee
  - Texas Clinical Research Institute, Arlington, Texas
  - Dallas Diabetes and Endocrine Center, Dallas, Texas
  - American Research Corporation at Texas Liver Institute, San Antonio, Texas
  - Clinical Trials of Texas, San Antonio, Texas
  - Endeavor Clinical Trials, San Antonio, Texas
  - Pioneer Research Solutions, Sugar Land, Texas
- Novartis Investigative Site, San Juan Bautista, Buenos Aires, Argentina
- Novartis Investigative Site, Mechelen, Belgium
- Brazil (3):
  - Novartis Investigative Site, Salvador, Estado de Bahia
  - Novartis Investigative Site, Porto Alegre, Rio Grande do Sul
  - Novartis Investigative Site, São Paulo, São Paulo
- Novartis Investigative Site, Sofia, Bulgaria
- Novartis Investigative Site, Montreal, Quebec, Canada
- Chile (2):
  - Novartis Investigative Site, Valdivia, Los Ríos Region
  - Novartis Investigative Site, Viña del Mar, Región de Valparaíso
- Colombia (3):
  - Novartis Investigative Site, Medellín, Antioquia
  - Novartis Investigative Site, Rionegro, Antioquia
  - Novartis Investigative Site, Bogotá
- Novartis Investigative Site, Aarhus N, Denmark
- Novartis Investigative Site, Tallinn, Estonia
- Germany (4):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Mainz
- Novartis Investigative Site, New Delhi, National Capital Territory of Delhi, India
- Italy (4):
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Rozzano, MI
  - Novartis Investigative Site, Palermo, PA
  - Novartis Investigative Site, Padua, PD
- Japan (4):
  - Novartis Investigative Site, Takamatsu, Kagawa-ken
  - Novartis Investigative Site, Yokohama, Kanagawa
  - Novartis Investigative Site, Saga, Saga-ken
  - Novartis Investigative Site, Izumo, Shimane
- Mexico (4):
  - Novartis Investigative Site, Guadalajara, Jalisco
  - Novartis Investigative Site, Cuauhtémoc, Mexico City
  - Novartis Investigative Site, Monterrey, Nuevo León
  - Novartis Investigative Site, México
- FDI Clinical Research, San Juan, Puerto Rico
- Russia (3):
  - Novartis Investigative Site, Novosibirsk
  - Novartis Investigative Site, Saint Petersburg
  - Novartis Investigative Site, Samara
- Novartis Investigative Site, Singapore, Singapore
- South Africa (2):
  - Novartis Investigative Site, Port Elizabeth, Eastern Cape
  - Novartis Investigative Site, Cape Town
- South Korea (2):
  - Novartis Investigative Site, Dongjak Gu, Seoul
  - Novartis Investigative Site, Seoul
- Spain (2):
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Madrid
- Taiwan (2):
  - Novartis Investigative Site, Kaohsiung City
  - Novartis Investigative Site, Tainan
- Novartis Investigative Site, Istanbul, Topkapi, Turkey (Türkiye)
- United Kingdom (2):
  - Novartis Investigative Site, Aberdeen, Grampian Region
  - Novartis Investigative Site, London

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing access to patient-level data and supporting clinical documents from eligible studies with qualified external researchers. Requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to protect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 234 participants were randomized at 81 sites.
Pre-assignment Details: One of the randomized participants in the tropifexor group was not treated due to loss of interest in the study.
Groups:
- Tropifexor Monotherapy: Tropifexor monotherapy arm: tropifexor 140 mcg capsule (+ placebo matching licogliflozin tablet), once daily orally
- Licogliflozin Monotherapy: Licogliflozin monotherapy arm: licogliflozin 30 mg tablet (+ placebo matching tropifexor capsule), once daily orally
- Combination Therapy: Combination therapy arm: tropifexor 140 mcg capsule + licogliflozin 30 mg tablet, once daily orally
- Placebo: Placebo arm: placebo matching tropifexor capsule + placebo matching licogliflozin tablet, once daily
Period: Overall Study
Arm/Group | Tropifexor Monotherapy | Licogliflozin Monotherapy | Combination Therapy | Placebo
Started | 54 | 55 | 84 | 41
Completed | 25 | 33 | 42 | 21
Not Completed | 29 | 22 | 42 | 20
Not completed — Adverse Event | 4 | 2 | 10 | 1
Not completed — Lost to Follow-up | 1 | 2 | 2 | 2
Not completed — Physician Decision | 1 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 1 | 0 | 0
Not completed — Study terminated by Sponsor | 22 | 16 | 28 | 17
Not completed — Withdrawal by Subject | 1 | 1 | 2 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS): all participants to whom study treatment was assigned by randomization and were treated
Groups:
- Total: Total of all reporting groups
Arm/Group | Tropifexor Monotherapy | Licogliflozin Monotherapy | Combination Therapy | Placebo | Total
Number analyzed (Participants) | 53 | 55 | 84 | 41 | 233
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 42 | 39 | 70 | 35 | 186
  >=65 years | 11 | 16 | 14 | 6 | 47
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.5 (11.09) | 56.0 (12.13) | 54.7 (10.82) | 54.9 (10.22) | 55.0 (11.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 34 | 43 | 26 | 129
  Male | 27 | 21 | 41 | 15 | 104
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 39 | 40 | 63 | 32 | 174
  Black or African American | 0 | 4 | 3 | 0 | 7
  Asian | 9 | 10 | 17 | 5 | 41
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 0 | 1
  American Indian or Alaska Native | 4 | 0 | 0 | 4 | 8
  Unknown | 0 | 1 | 1 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Histological Improvement: Number and Percentage of Participants Who Responded at Week 48 Compared With Baseline
Description: Response was defined as at least a one-stage improvement in fibrosis without worsening of nonalcoholic steatohepatitis (NASH)
  Fibrosis staging and Nonalcoholic Fatty Liver Disease (NAFLD) Activity Score (NAS) based on steatosis, lobular inflammation, and hepatocyte ballooning assessment were determined by a Study Central Reader. NASH CRN fibrosis criteria: Stage 0 = no fibrosis; Stage 1 = centrilobular pericellular fibrosis (or periportal fibrosis in children); Stage 2 = centrilobular and periportal fibrosis; Stage 3 = bridging fibrosis; and Stage 4 = cirrhosis.
Time Frame: Baseline, Week 48
Population: Full Analysis Set (FAS): all participants to whom study treatment has been assigned by randomization and had an assessment of response at Week 48. Efficacy analysis was conducted using the FAS.
Measure: Count of Participants; unit: Participants
Arm/Group | Tropifexor Monotherapy | Licogliflozin Monotherapy | Combination Therapy | Placebo
Number analyzed (Participants) | 23 | 28 | 34 | 17
Participants | 6 | 9 | 10 | 4

2. Primary Outcome: Number and Percentage of Participants With Resolution of NASH and no Worsening of Fibrosis
Description: Fibrosis staging and Nonalcoholic Fatty Liver Disease (NAFLD) Activity Score (NAS) based on steatosis, lobular inflammation, and hepatocyte ballooning assessment were determined by a Study Central Reader. NASH CRN fibrosis criteria: Stage 0 = no fibrosis; Stage 1 = centrilobular pericellular fibrosis (or periportal fibrosis in children); Stage 2 = centrilobular and periportal fibrosis; Stage 3 = bridging fibrosis; and Stage 4 = cirrhosis.
Time Frame: 48 weeks
Population: Full Analysis Set (FAS): all participants to whom study treatment has been assigned by randomization. Efficacy analysis was conducted using the FAS
Measure: Count of Participants; unit: Participants
Arm/Group | Tropifexor Monotherapy | Licogliflozin Monotherapy | Combination Therapy | Placebo
Number analyzed (Participants) | 23 | 28 | 34 | 17
Participants | 5 | 3 | 10 | 2

3. Secondary Outcome: Number and Percentage of Participants Who Achieved Resolution of NASH and no Worsening of Fibrosis OR Improvement in Fibrosis by at Least One Stage Without Worsening of NASH
Description: as for outcome 2
Time Frame: 48 weeks
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | Tropifexor Monotherapy | Licogliflozin Monotherapy | Combination Therapy | Placebo
Number analyzed (Participants) | 23 | 28 | 34 | 17
Participants | 8 | 10 | 14 | 5

4. Secondary Outcome: Number and Percentage of Participants With at Least One Stage Improvement in Fibrosis
Description: as for outcome 2
Time Frame: 48 weeks
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | Tropifexor Monotherapy | Licogliflozin Monotherapy | Combination Therapy | Placebo
Number analyzed (Participants) | 23 | 28 | 34 | 17
Participants | 6 | 10 | 11 | 4

5. Secondary Outcome: Number and Percentage of Participants With at Least Two Stage Improvement in Fibrosis Without Worsening of NASH
Description: Fibrosis staging and Non-alcoholic Fatty Liver Disease (NAFLD) Activity Score (NAS) based on steatosis, lobular inflammation, and hepatocyte ballooning assessment were determined by a Study Central Reader. NASH CRN fibrosis criteria: Stage 0 = no fibrosis; Stage 1 = centrilobular pericellular fibrosis (or periportal fibrosis in children); Stage 2 = centrilobular and periportal fibrosis; Stage 3 = bridging fibrosis; and Stage 4 = cirrhosis.
Time Frame: 48 weeks
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | Tropifexor Monotherapy | Licogliflozin Monotherapy | Combination Therapy | Placebo
Number analyzed (Participants) | 23 | 28 | 34 | 17
Participants | 3 | 4 | 3 | 3

6. Secondary Outcome: Number and Percentage of Participants Achieving 5% or More Reduction in Body Weight at Week 48 Compared With Baseline
Description: Whether the participants had 5% or more reduction in body weight.
Time Frame: Baseline, Week 48
Population: Data are reported for the total number of participants in the treatment group with response variable defined.
Measure: Count of Participants; unit: Participants
Arm/Group | Tropifexor Monotherapy | Licogliflozin Monotherapy | Combination Therapy | Placebo
Number analyzed (Participants) | 23 | 32 | 35 | 24
Participants | 12 | 9 | 28 | 3

7. Secondary Outcome: Change From Baseline to Week 48 in Percent Liver Fat Content Based on Magnetic Resonance Imaging - Proton Density Fat Fraction (MRI - PDFF)
Description: Change in liver fat content based on MRI-PDFF.
Time Frame: Baseline, Week 48
Population: FAS: all participants to whom study treatment has been assigned by randomization and had an assessment at Week 48. This analysis was performed in 40% of participants.
Measure: Mean (Standard Deviation); unit: Percent liver fat
Arm/Group | Tropifexor Monotherapy | Licogliflozin Monotherapy | Combination Therapy | Placebo
Number analyzed (Participants) | 15 | 19 | 21 | 20
Percent liver fat | -6.57 (5.913) | -2.64 (5.866) | -7.69 (6.702) | -2.58 (3.599)

8. Secondary Outcome: Change From Baseline in Alanine Transaminase (ALT) Over Time
Description: To determine the relationship of investigational treatment and markers of hepatic inflammation in NASH.
Time Frame: Baseline to Weeks 2, 4, 8, 12, 16, 20, 24, 32, 40, 48, follow-up (up to 62 weeks)
Population: The safety analysis set included all participants who received at least one dose of study treatment. At each time point, only participants with a value at both Baseline and that time point were included.
Measure: Mean (Standard Deviation); unit: units per liter (U/L)
Arm/Group | Tropifexor Monotherapy | Licogliflozin Monotherapy | Combination Therapy | Placebo
Number analyzed (Participants) | 53 | 55 | 84 | 41
units per liter (U/L)
  Week 2: number analyzed (Participants) | 50 | 51 | 79 | 38
  Week 2 | -17.4 (28.30) | -3.2 (15.52) | -13.5 (24.47) | -4.3 (18.94)
  Week 4: number analyzed (Participants) | 50 | 50 | 75 | 40
  Week 4 | -16.1 (18.41) | -4.2 (19.84) | -14.5 (25.78) | -3.2 (17.81)
  Week 8: number analyzed (Participants) | 47 | 51 | 64 | 39
  Week 8 | -9.9 (20.02) | -7.9 (19.82) | -17.6 (23.47) | -5.6 (19.67)
  Week 12: number analyzed (Participants) | 47 | 46 | 59 | 38
  Week 12 | -13.8 (28.48) | -11.3 (16.57) | -21.0 (24.91) | -2.5 (25.05)
  Week 16: number analyzed (Participants) | 39 | 47 | 54 | 35
  Week 16 | -15.4 (26.94) | -12.4 (20.38) | -24.4 (26.13) | -3.2 (24.57)
  Week 20: number analyzed (Participants) | 41 | 43 | 52 | 34
  Week 20 | -14.5 (27.92) | -14.6 (24.96) | -25.0 (28.95) | -5.7 (20.20)
  Week 24: number analyzed (Participants) | 40 | 38 | 42 | 35
  Week 24 | -15.1 (28.34) | -17.0 (22.43) | -35.2 (30.61) | -4.0 (28.28)
  Week 32: number analyzed (Participants) | 37 | 36 | 44 | 28
  Week 32 | -18.2 (30.97) | -13.0 (28.01) | -33.8 (37.21) | -1.0 (41.32)
  Week 40: number analyzed (Participants) | 28 | 34 | 37 | 29
  Week 40 | -12.7 (39.35) | -15.2 (26.91) | -36.1 (27.42) | -8.7 (40.70)
  Week 48: number analyzed (Participants) | 22 | 32 | 33 | 21
  Week 48 | -11.7 (49.32) | -12.0 (28.99) | -36.9 (30.20) | -19.5 (30.16)
  Follow-up: number analyzed (Participants) | 45 | 49 | 75 | 34
  Follow-up | -1.5 (37.77) | -9.4 (27.94) | -17.0 (27.97) | -8.8 (28.88)

9. Secondary Outcome: Change From Baseline in Aspartate Aminotransferase (AST) Over Time
Description: To determine the relationship of investigational treatment and markers of hepatic inflammation in NASH.
Time Frame: Baseline to Weeks 2, 4, 8, 12, 16, 20, 24, 32, 40, 48, follow-up (up to 62 weeks)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Tropifexor Monotherapy | Licogliflozin Monotherapy | Combination Therapy | Placebo
Number analyzed (Participants) | 53 | 55 | 84 | 41
U/L
  Week 2: number analyzed (Participants) | 50 | 51 | 81 | 40
  Week 2 | -7.9 (14.93) | -3.9 (12.98) | -5.5 (19.38) | -1.8 (13.46)
  Week 4: number analyzed (Participants) | 50 | 52 | 75 | 40
  Week 4 | -1.7 (17.43) | -2.4 (20.49) | -4.9 (22.19) | -2.2 (15.35)
  Week 8: number analyzed (Participants) | 50 | 52 | 66 | 39
  Week 8 | 1.2 (23.71) | -7.4 (14.12) | -6.7 (20.13) | -1.6 (15.19)
  Week 12: number analyzed (Participants) | 47 | 47 | 60 | 38
  Week 12 | 0.4 (21.34) | -10.3 (13.25) | -10.4 (21.42) | -1.4 (19.08)
  Week 16: number analyzed (Participants) | 41 | 48 | 55 | 35
  Week 16 | -0.7 (21.71) | -10.8 (16.37) | -12.9 (20.98) | -2.4 (17.42)
  Week 20: number analyzed (Participants) | 42 | 43 | 51 | 35
  Week 20 | -1.0 (22.46) | -10.0 (19.81) | -10.8 (25.98) | -3.9 (14.23)
  Week 24: number analyzed (Participants) | 40 | 38 | 44 | 35
  Week 24 | -1.4 (19.96) | -13.8 (19.81) | -18.3 (23.26) | -2.2 (21.96)
  Week 32: number analyzed (Participants) | 37 | 37 | 44 | 30
  Week 32 | -2.0 (32.00) | -11.2 (20.12) | -15.4 (34.92) | -1.1 (29.62)
  Week 40: number analyzed (Participants) | 28 | 34 | 36 | 30
  Week 40 | 3.2 (34.40) | -11.9 (20.22) | -20.6 (22.57) | -5.9 (23.21)
  Week 48: number analyzed (Participants) | 23 | 31 | 34 | 24
  Week 48 | -0.7 (31.34) | -11.3 (23.53) | -20.4 (24.19) | -12.8 (17.01)
  Follow-up: number analyzed (Participants) | 47 | 48 | 77 | 35
  Follow-up | -2.0 (21.21) | -8.2 (24.01) | -10.6 (21.27) | -3.3 (23.64)

10. Secondary Outcome: Change From Baseline in Gamma-glutamyltransferase (GGT) Over Time
Description: To determine the relationship of investigational treatment and markers of hepatic inflammation in NASH.
Time Frame: Baseline to Weeks 2, 4, 8, 12, 16, 20, 24, 32, 40, 48, follow-up (up to 62 weeks)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Tropifexor Monotherapy | Licogliflozin Monotherapy | Combination Therapy | Placebo
Number analyzed (Participants) | 53 | 55 | 84 | 41
U/L
  Week 2: number analyzed (Participants) | 50 | 52 | 81 | 39
  Week 2 | -34.8 (46.06) | -2.8 (21.81) | -30.6 (45.85) | 3.8 (34.60)
  Week 4: number analyzed (Participants) | 50 | 52 | 75 | 40
  Week 4 | -43.6 (60.28) | -7.0 (20.56) | -41.7 (60.81) | -1.1 (31.63)
  Week 8: number analyzed (Participants) | 49 | 52 | 66 | 40
  Week 8 | -37.9 (37.85) | -15.3 (28.06) | -45.0 (69.45) | -0.9 (33.16)
  Week 12: number analyzed (Participants) | 47 | 46 | 60 | 38
  Week 12 | -37.4 (96.36) | -17.5 (33.83) | -48.0 (76.04) | 5.2 (25.03)
  Week 16: number analyzed (Participants) | 41 | 48 | 54 | 35
  Week 16 | -39.4 (41.77) | -15.5 (33.94) | -52.2 (78.29) | 2.2 (36.71)
  Week 20: number analyzed (Participants) | 42 | 44 | 52 | 35
  Week 20 | -32.9 (37.55) | -14.8 (41.11) | -50.1 (79.30) | -0.8 (45.84)
  Week 24: number analyzed (Participants) | 40 | 38 | 44 | 35
  Week 24 | -32.0 (45.55) | -22.3 (28.06) | -58.1 (82.45) | 3.3 (44.08)
  Week 32: number analyzed (Participants) | 37 | 36 | 44 | 29
  Week 32 | -34.5 (37.31) | -19.4 (28.68) | -55.1 (76.85) | 8.2 (45.21)
  Week 40: number analyzed (Participants) | 28 | 34 | 37 | 30
  Week 40 | -38.8 (42.89) | -20.6 (30.99) | -50.0 (72.08) | 0.2 (54.04)
  Week 48: number analyzed (Participants) | 23 | 32 | 34 | 24
  Week 48 | -31.6 (46.00) | -20.1 (29.10) | -44.1 (67.27) | -11.1 (38.01)
  Follow-up: number analyzed (Participants) | 47 | 49 | 77 | 35
  Follow-up | 14.8 (69.63) | -9.4 (42.96) | 5.6 (139.33) | 7.3 (43.69)

ADVERSE EVENTS:
Time Frame: Up to approximately 52 weeks
Description: An AE is any untoward medical occurrence, unfavorable, or unintended sign (including an abnormal laboratory finding), symptom, disease, or injury, that ocurred during treatment period. They include events that started after the first dose of study treatment or events that were present prior to start of study treatment but increased in severity during on-treatment period. The safety analysis set included all participants who received at least one dose of study treatment.
Groups:
- LJN452: Tropifexor monotherapy arm: tropifexor 140 mcgcapsule (+ placebo matching licogliflozin tablet), once daily orally
- LIK066: Licogliflozin monotherapy arm: licogliflozin 30 mg tablet (+ placebo matching tropifexor capsule), once daily orally
- Combination: Combination therapy arm: tropifexor 140 mcg capsule + licogliflozin 30 mg tablet, once daily orally
- All Patients: All Patients
Arm/Group | LJN452 | LIK066 | Combination | Placebo | All Patients
All-Cause Mortality (participants affected / at risk) | 0/53 | 0/55 | 0/84 | 0/41 | 0/233
Serious Adverse Events (participants affected / at risk) | 4/53 | 3/55 | 4/84 | 3/41 | 14/233
Other Adverse Events (participants affected / at risk) | 35/53 | 39/55 | 54/84 | 23/41 | 151/233
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LJN452 (N=53) | LIK066 (N=55) | Combination (N=84) | Placebo (N=41) | All Patients (N=233)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1 | 1
Cardiac failure chronic (Cardiac disorders) | 1 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Haemoperitoneum (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 1 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 1
Haemobilia (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 1
COVID-19 pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Hepatitis E (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Post procedural fever (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 1
Sciatica (Nervous system disorders) | 0 | 0 | 1 | 0 | 1
Calculus urinary (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LJN452 (N=53) | LIK066 (N=55) | Combination (N=84) | Placebo (N=41) | All Patients (N=233)
Abdominal distension (Gastrointestinal disorders) | 2 | 3 | 5 | 2 | 12
Abdominal pain upper (Gastrointestinal disorders) | 4 | 2 | 1 | 1 | 8
Diarrhoea (Gastrointestinal disorders) | 7 | 21 | 21 | 6 | 55
Dyspepsia (Gastrointestinal disorders) | 2 | 4 | 2 | 1 | 9
Flatulence (Gastrointestinal disorders) | 4 | 4 | 3 | 0 | 11
Nausea (Gastrointestinal disorders) | 6 | 4 | 7 | 2 | 19
Vomiting (Gastrointestinal disorders) | 7 | 2 | 3 | 2 | 14
Fatigue (General disorders) | 3 | 0 | 1 | 1 | 5
Pyrexia (General disorders) | 0 | 5 | 0 | 1 | 6
COVID-19 (Infections and infestations) | 1 | 10 | 9 | 9 | 29
Urinary tract infection (Infections and infestations) | 3 | 6 | 4 | 2 | 15
Glucose urine present (Investigations) | 2 | 3 | 2 | 0 | 7
Urine albumin/creatinine ratio increased (Investigations) | 1 | 2 | 2 | 3 | 8
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 3 | 6
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 3 | 2 | 1 | 6
Dizziness (Nervous system disorders) | 3 | 2 | 2 | 0 | 7
Headache (Nervous system disorders) | 2 | 1 | 3 | 6 | 12
Insomnia (Psychiatric disorders) | 4 | 0 | 1 | 0 | 5
Haematuria (Renal and urinary disorders) | 0 | 3 | 0 | 0 | 3
Balanoposthitis (Reproductive system and breast disorders) | 0 | 4 | 1 | 0 | 5
Pruritus (Skin and subcutaneous tissue disorders) | 20 | 9 | 22 | 4 | 55
Rash (Skin and subcutaneous tissue disorders) | 2 | 3 | 0 | 2 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2021-04-30): https://cdn.clinicaltrials.gov/large-docs/41/NCT04065841/Prot_000.pdf
  • Statistical Analysis Plan (2019-12-09): https://cdn.clinicaltrials.gov/large-docs/41/NCT04065841/SAP_001.pdf